CLINICAL TRIAL: NCT07012811
Title: Evaluation of Topical Tretinoin 0.05% Alone Versus Combination With Oral Isotretinoin (0.5 mg/kg/Day) in the Treatment of Plane Warts
Brief Title: Treatment of Plane Warts With Topical and Oral Retinoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TishreenU - Plane Warts
Record Dates: First submitted 2025-05-29; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Plane Warts
Keywords: Human papillomavirus; Tretinoin; Isotretinoin
MeSH Terms: interventions — Tretinoin; Isotretinoin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients apply tretinoin cream 0.05% once daily at night for 3 months
  Interventions: Drug: Topical tretinoin 0.05%
- Group B (Experimental): Patients apply tretinoin cream 0.05% and receive oral isotretinoin capsule in the dose of 0.5 mg/kg/day for 3 months
  Interventions: Drug: Topical tretinoin 0.05% + oral isotretinoin (0.5 mg/kg/day)

INTERVENTIONS:
Drug: Topical tretinoin 0.05% — Topical tretinoin cream 0.05% applied once daily at night
  Arms: Group A
Drug: Topical tretinoin 0.05% + oral isotretinoin (0.5 mg/kg/day) — Topical tretinoin cream 0.05% once daily at night + oral isotretinoin capsule in the dose of 0.5 mg/kg/day
  Arms: Group B

SUMMARY:
The aim of this study was to compare the effectiveness and safety of topical tretinoin cream 0.05% alone against combination with oral isotretinoin (0.5 mg/kg/day) for treatment of plane warts.

DETAILED DESCRIPTION:
This study included 39 patients divided into two groups. Treatment was given for three months duration. Patients were followed-up for further three months to assess the recurrence rate. Combination treatment led to a faster resolution and a higher percentage of complete response. It presents a promising effective alternative option for treatment of plane warts.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 12 years diagnosed with plane warts.
* Patients who had not received any treatment for warts in the last month.

Exclusion Criteria:

* Pregnancy and lactation.
* Abnormal lipid profile.
* Significant hepatic or renal dysfunction.
* Depression.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Response Rate, as Measured by the Reduction in Number of Lesions at Week 4 | Week 4
  The response is assessed according to the decrease in number of lesions as followed: complete response (total clearance of warts), partial response (decease in the number of lesion ≥ 50%), no response (decrease in the number of lesion <50% or no clearance).
Response Rate, as Measured by the Reduction in Number of Lesions at Week 8 | Week 8
  The response is assessed according to the decrease in number of lesions as followed: complete response (total clearance of warts), partial response (decease in the number of lesion ≥ 50%), no response (decrease in the number of lesion <50% or no clearance).
Response Rate, as Measured by the Reduction in Number of Lesions at Week 12 | Week 12
  The response is assessed according to the decrease in number of lesions as followed: complete response (total clearance of warts), partial response (decease in the number of lesion ≥ 50%), no response (decrease in the number of lesion <50% or no clearance).

SECONDARY OUTCOMES:
Safety, as Measured by the Number of Patients With at Least one Adverse Effect | week 12
  The adverse effects are defined as unwanted effects related directly to the drug
Recurrence Rate, as Measured by the Number of Patients who Have Recurrent Lesions After 12 Weeks of Termination of Therapy | 12 weeks after termination of therapy
  The recurrence is defined as reappearance of lesions at the same locations after complete response

CONTACTS AND LOCATIONS:
Overall Officials: Zeina M Habib, MD, Principal Investigator — Tishreen University Hospital
Locations (1):
- Tishreen University- Faculty of Medicine, Latakia, Latakia Governorate, Syria

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of this study after deidentification
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 2 months and ending 5 months following publication
Access Criteria: researchers who provide a methodological proposal

REFERENCES:
- [Background] Singh R, Pandey SS: Efficacy of topical 5% 5-fluorouracil and 0.05% tretinoin and electrosurgery in the treatment of plane warts: a randomized controlled comparative trial. Nepal J Dermatol Venereol & Leprol. 2021, 19(1):55-9
- [Background] Randhawa NK, Kumar S, Agarwal US, Agarwal P, Bansal A, Meena S: To evaluate efficacy and safety of low dose oral isotretinoin (20 mg/day) alone versus combination of low dose oral isotretinoin (20 mg/day) plus topical tretinoin (0.1%) in gel formulation in the treatment of verruca plana. J Clin Exp Dermatol Res. 2023, 14:635.
- [Background] Nooruldeen AD, Saeed MY: Efficacy and safety of oral isotretinoin in treatment of plane warts. Bali Med J. 2021, 10(3): 1076-7080
- [Background] Dong ZY, He MJ, Hu Y, Wang F, Ran DL, Fu DS, He Q, Yang RP, Zhang JA. Unveiling the Mechanism of Retinoic Acid Therapy for Cutaneous Warts: Insights from Multi-Omics Integration. Clin Cosmet Investig Dermatol. 2024 Dec 18;17:2923-2932. doi: 10.2147/CCID.S504391. eCollection 2024. PMID 39712939
- [Background] Kaur GJ, Brar BK, Kumar S, Brar SK, Singh B. Evaluation of the efficacy and safety of oral isotretinoin versus topical isotretinoin in the treatment of plane warts: a randomized open trial. Int J Dermatol. 2017 Dec;56(12):1352-1358. doi: 10.1111/ijd.13727. Epub 2017 Sep 13. PMID 28901534
- [Background] Sterling JC, Gibbs S, Haque Hussain SS, Mohd Mustapa MF, Handfield-Jones SE. British Association of Dermatologists' guidelines for the management of cutaneous warts 2014. Br J Dermatol. 2014 Oct;171(4):696-712. doi: 10.1111/bjd.13310. Epub 2014 Oct 1. No abstract available. PMID 25273231